CLINICAL TRIAL: NCT06129370
Title: Testing of a Medication Dosing Software for Pediatric Emergency Care
Brief Title: Testing of Medication Dosing Software
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nura Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2024-10183
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Emergency Medicine
Keywords: Simulation; Pediatric emergency care; Healthcare professionals; Medication errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Software, then Standard (Experimental): Participants will use the medication dosage software to calculate and prepare intravenous medications during the initial run through of pediatric case scenarios. Then, they will use standard clinical practice (Lexicomp and manual calculator) during the second run through of pediatric case scenarios.
  Interventions: Device: Standard practice; Device: Medication dosing software
- Standard, then Software (Experimental): Participants will use standard clinical practice (Lexicomp and manual calculator) to calculate and prepare intravenous medications during the initial run through of pediatric case scenarios. Then, they will use the medication dosage software during the second run through of pediatric case scenarios.
  Interventions: Device: Standard practice; Device: Medication dosing software

INTERVENTIONS:
Device: Standard practice — Lexicomp and manual calculator
Device: Medication dosing software — Medication dosing software

SUMMARY:
The goal of this clinical study is to evaluate the clinical efficiency of a medication dosing software in simulated pediatric emergency care. The main questions it aims to answer are:

* Will the time to patient be significantly reduced with the medication dosage software when compared to standard clinical practice?
* Will the time to calculate dosage of medications be significantly reduced with the medication dosage software when compared to standard clinical practice?
* How will users perceive clinical efficiency, ease of use, confidence level of using the medication dosage software when compared to standard clinical practice?
* How will accuracy of medication dose and volume calculations as well as final volume ready for administration using the medication dosage software compared to standard clinical practice?
* Will the time spent calculating medication doses by the second healthcare professional on pediatric non-acute and acute care cases be significantly reduced with the medication dosage software when compared to standard clinical practice?

Participants will be presented pediatric care scenarios and asked to calculate and prepare intravenous medications under two interventions: the medication dosage software and standard clinical practice (Lexicomp and manual calculator).

ELIGIBILITY:
Inclusion Criteria:

-Healthcare professionals who have worked or who are currently working at a healthcare facility and involved in the calculation or preparation of IV medication.

Exclusion Criteria:

* Healthcare professionals who cannot read, speak, or understand English or French as the simulations will be conducted in English or French.
* Performance of physically strenuous activity 30 min prior to study.
* Physical limitations that affect performance on required tasks (e.g., inability to place arm cuff on mannequin's arm, inability to handle weight estimation and touchscreen devices).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
TIme to patient | Through study completion, up to 3 months
  Assess the time elapsed from ordering of medication to ready for administration using the medication dosage software compared to the time achieved with standard clinical practice
Time to calculate | Through study completion, up to 3 months
  Assess the time to calculate medication dosage using the medication dosage software compared to standard clinical practice

SECONDARY OUTCOMES:
Feedback | Through study completion, up to 3 months
  time to calculate medication dosage using the medication dosage software compared to standard clinical practice
Accuracy | Through study completion, up to 3 months
  To assess the accuracy of (I) medication dose and volume calculations and (II) final volume ready for administration using the medication dosage software compared to standard clinical practice.
Time of calculation by second healthcare professional | Through study completion, up to 3 months
  To assess the time spent calculating medication dosages by the second healthcare professional.

IPD SHARING:
Plan to Share IPD: Undecided